CLINICAL TRIAL: NCT06215664
Title: A Randomized Controlled Trial of a Game-Based Intervention to Reduce Alcohol-Related Harms Among Sexual and Gender Minority Youth
Brief Title: Game-Based Intervention to Reduce Alcohol-Related Harms Among Sexual and Gender Minority Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Coulter, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY23030071; R01AA030017 (NIH)
Record Dates: First submitted 2023-12-18; First posted 2024-01-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Problem; Harm Reduction; Alcohol-Related Harm
MeSH Terms: conditions — Alcohol-Related Disorders; Harm Reduction

STUDY DESIGN:
Intervention Model Description: Two-armed parallel randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Singularities Game (Experimental): Singularities is an online game.
  Interventions: Behavioral: Singularities Game
- Food4Thought (Active Comparator): Food4Thought is an attention control condition in which we provide participants with similar amounts of research team contact and program contact as the intervention. Participants will play the game Pick Your Plate! A Global Guide to Nutrition, developed by the Smithsonian Science Education Center. Participants are instructed to build healthy meals using cuisine from around the world while ensuring they stick to a budget and meet all their nutritional needs. Food4Thought will be delivered via Qualtrics.
  Interventions: Behavioral: Food4Thought

INTERVENTIONS:
Behavioral: Singularities Game — Singularities is a theory-based, community-informed, web-accessible, roleplaying game-based intervention incorporating 4 primary components: fostering healthy identity development in a safe environment; encouraging help-seeking behaviors; encouraging use of productive coping; alcohol-harm reduction; and encouraging healthy internet and social media use.
  Arms: Singularities Game
Behavioral: Food4Thought — Food4Thought is an attention control condition in which we provide participants with similar amounts of research team contact and program contact as the intervention. Participants will play the game Pick Your Plate! A Global Guide to Nutrition, developed by the Smithsonian Science Education Center. Participants are instructed to build healthy meals using cuisine from around the world while ensuring they stick to a budget and meet all their nutritional needs. Food4Thought will be delivered via Qualtrics.
  Arms: Food4Thought

SUMMARY:
This is a randomized controlled trial to examine the efficacy of a game-based intervention to reduce alcohol-related harms among sexual and gender minority youth.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in English
* Live in the U.S.,
* 14-18 years old
* Have a sexual minority identity (i.e., gay, lesbian, bisexual, or queer) or a gender minority identity (i.e., consider themselves to be transgender or nonbinary),
* Have an internet-accessible computer, smart phone, or tablet,
* Provide an email address.
* Have drank alcohol in their lifetime or intend to in the next year.

Exclusion Criteria:

* Cisgender heterosexuals.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Any gender minorities are eligible as are any cisgender sexual minority people.
Enrollment: 1992 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol-related harms | 3 months
  Primary outcome is alcohol-related harms defined as the frequency of 19 total harms (e.g., Hangover after drinking, Unable to remember what happened after drinking, Had sex that you later regretted, Trouble with parent(s) because of drinking Physical fight because you were affected by alcohol, Drove in a vehicle after drinking) as measured in the School Health and Alcohol Harm Reduction Project (SHAHRP)

SECONDARY OUTCOMES:
Drinking Quantity | 3 months
  Number of drinks consumed on a typical day of drinking in the past three months via Quantity-Frequency items
Drinking Frequency | 3 months
  Number of days on which one or more drinks were consumed in past month via Quantity-Frequency items.
Binge Drinking | 3 months
  Number of times where 4 or 5+ drinks (asking both, regardless of assigned/biological sex at birth to be inclusive of gender minorities) were consumed in a 2-hour period over the past 3 months, via NIAAA items
Alcohol Use Initiation | 3 months
  Survey item from the Youth Risk Behavior Survey assessing lifetime alcohol use.
Alcohol Harm Reduction Skills | 3 months
  Which behaviors are engaged in while drinking or partying, measured with the Protective Behavioral Strategies Scale (PBSS). Scores range from 20 to 120, with higher scores indicating more skills used
Bystander Alcohol Harm Reduction Skills | 3 months
  Total # of times a specific strategy was used to help others before, during, or after drinking, using the Strategies subscale of the Bystanders to Alcohol Risk Scale (BARS). Scores range from 0 to 27, with higher scores indicating more skills used
Emotional distress tolerance skills | 3 months
  Beliefs about feeling distressed or upset, measured with the Distress Tolerance Scale (DTS). Scores range from 15 to 75, with higher scores indicating a poorer outcome
Emotion regulation and decentering practices | 3 months
  How often mindfulness practices are used, measured with the Applied Mindfulness Process Scale (AMPS). Scores range from 0 to 60, with higher scores indicating a better outcome
Healthy social media use | 3 months
  Endorsement of beliefs and thoughts about social media, using MetroWest Adolescent Health Survey items

CONTACTS AND LOCATIONS:
Overall Officials: Robert WS Coulter, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan and archiving of de-identified data as required by NIH
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after end of study
Access Criteria: Public
URL: https://nda.nih.gov/niaaa